CLINICAL TRIAL: NCT00106262
Title: A Phase II Study of VELCADE TM(PS-341) and Irinotecan in the Treatment of Progressive, Recurrent or Metastatic Cervical, Vulvar, or Vaginal Cancer
Brief Title: Study of Velcade and Irinotecan in Advanced Cervical, Vulvar, or Vaginal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05122
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Cervical Cancer
Keywords: advanced cervical cancer; metastatic cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bortezomib; Irinotecan

INTERVENTIONS:
Drug: Velcade (bortezomib)
Drug: Irinotecan

SUMMARY:
This study is conducting an evaluation of two chemotherapy drugs, Velcade and Irinotecan, in women with advanced, recurrent, or metastatic cervical cancer, vaginal cancer, or vulvar cancer. Patients with cervical cancer may have received a platinum-containing treatment as systemic therapy without radiation, but is not required.

DETAILED DESCRIPTION:
This is a phase 2 study. Patients with advanced or metastatic histologically documented squamous cell carcinoma, adenocarcinoma, or adenosquamous cancers originating in the cervix, vagina, or vulva will be eligible. Measurable disease by either clinical exam or radiography is also required. Patients receiving cisplatin-based chemoradiation as definitive treatment for local disease will be eligible. Patients must have no more than one prior platinum-based chemotherapy regimen in the metastatic setting. Patients presenting with distant metastatic disease (beyond the pelvis) will be eligible, as long as they are not eligible for a higher priority study.

ELIGIBILITY:
Inclusion Criteria

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* age > 18
* Karnofsky performance status > 60%
* Measurable disease on clinical exam or by RECIST criteria
* One prior platinum-based systemic chemotherapy regimen for advanced disease is allowed but not required. Chemotherapy administered as a radiosensitizer in conjunction with primary radiotherapy is not considered a systemic chemotherapy regimen and is also allowed. Patients eligible for a higher priority study will be excluded.
* Life expectancy > 6 weeks
* Peripheral neuropathy ≤ Grade 2 by CTC 3.0 criteria
* Women of child-bearing potential must have a negative pregnancy test
* Adequate hematopoietic function defined as: ANC ≥ 1500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 8 g/dL.
* Adequate renal and hepatic function defined as: Bilirubin ≤ 1.5 times upper limit of normal (ULN); SGOT ≤ 2.5 times ULN; Alkaline phosphatase ≤ 2.5 times ULN; Creatinine ≤ 2 times ULN.

Exclusion Criteria

* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Prior treatment with CAMPTOSAR or VELCADE
* More than one prior treatment for metastatic disease.
* Concurrent uncontrolled illness
* Ongoing or active infection
* History or active secondary cancer within the last 5 years, except for superficial basal cell skin cancers
* Psychiatric illness or social situation that would preclude study compliance.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2005-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
overall response rate
time to progression

SECONDARY OUTCOMES:
overall survival
toxicity of this combination in women with advanced cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: Don S Dizon, MD, Principal Investigator — Women & Infants' Hospital of Rhode Island
Locations (1):
- Women & Infants' Hospital, Providence, Rhode Island, United States